CLINICAL TRIAL: NCT07311330
Title: A Randomized, Double-blind, Placebo-controlled Phase IIa Clinical Trial to Evaluate the Efficacy and Safety of YN001 in Patients With Atherosclerotic Cardiovascular and Cerebrovascular Diseases and Erectile Dysfunction
Brief Title: Phase IIa Clinical Trial of YN001 in Patients With Atherosclerotic Cardiovascular and Cerebrovascular Diseases and Erectile Dysfunction
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Inno Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YN001-006
Record Dates: First submitted 2025-11-19; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Atherosclerotic Cardiovascular Disease (ASCVD); Erectile Dysfunction
MeSH Terms: conditions — Atherosclerosis; Erectile Dysfunction | interventions — Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- YN001 20mg Dose + 5% glucose injection (Active Comparator): Specified dose on specified Days
  Interventions: Drug: YN001 20mg Dose + 5% glucose injection
- 5% glucose injection (Placebo Comparator): Specified dose on specified Days
  Interventions: Other: 5% glucose injection

INTERVENTIONS:
Drug: YN001 20mg Dose + 5% glucose injection — The treamtment group was given YN001 20 mg, once a week (QW), cumulative administration for 12 weeks (about 3 months)
  Arms: YN001 20mg Dose + 5% glucose injection
Other: 5% glucose injection — The control group was given placebo once a week (QW), cumulative administration for 12 weeks (about 3 months)
  Arms: 5% glucose injection

SUMMARY:
This is a randomized, double-blind, placebo-controlled phase IIa clinical trial to evaluate the efficacy and safety of YN001 in patients with atherosclerotic cardiovascular and cerebrovascular diseases and erectile dysfunction

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand the purpose, nature, method and possible adverse reactions of the study, voluntarily participate as a subject in the study, and sign the informed consent form (ICF) before performing any study-related assessments;
2. One or both of the previous history of coronary atherosclerosis, coronary heart disease, cerebral atherosclerosis, stroke, ischemic attack, carotid atherosclerosis, peripheral arterial disease, or plaque in at least one vessel of the carotid, subclavian, or femoral arteries as detected by peripheral arterial ultrasound .
3. Clinical diagnosis of mild to moderate erectile dysfunction, IIEF-5 questionnaire score ≤ 21 points, duration of at least 3 months (subject to signing informed consent);
4. Subjects (including partners) guarantee that they have no plans to father a child or donate sperm during the study and for 3 months after the last dose and voluntarily take appropriate contraceptive measures;
5. After the screening run-in period, the following three conditions were met simultaneously:

1) At least 4 attempts at sexual intercourse during the run-in period; 2) Has a failure rate of ≥ 50% of attempts to intercourse (failure to intercourse is defined as having at least one of the three questions answered on the SEP); 3) IIEF-EF score ≥ 11 and ≤ 25.

Exclusion Criteria:

1. Patients with erectile dysfunction caused by other sexual dysfunction diseases (such as ejaculatory dysfunction) or endocrine diseases that are not controlled (after medication) (such as hypogonadism, hyperthyroidism/hypothyroidism, pituitary tumor, etc.);
2. History of stroke within 6 months prior to informed consent;
3. Patients who have received or are receiving anti-androgen therapy, or have a history of androgen replacement therapy and are stable for less than 3 months;
4. Patients scheduled for CABG, PCI, heart transplantation, SAVR/TAVR during the study period;
5. Patients with unstable diabetic blood glucose control, and fasting blood glucose more than 15 mmol/L, or accompanied by diabetic complications (diabetic nephropathy, peripheral neuropathy);
6. Combined with abnormal liver function, defined as AST and/or ALT more than 2 times the upper limit of normal;
7. Combined with severe renal dysfunction, defined as glomerular filtration rate < 30.0 mL/min/1.73m ² calculated by CKD-EPI formula;
8. Subjects who have used vacuum aspiration (VCD), intracavernosal injection (ICI) therapy or other drugs to treat erectile dysfunction and cannot interrupt the above treatment during the study;
9. Patients who have severe central nervous system injury (cerebral vascular diseases such as cerebral hemorrhage or ischemia, brain inflammatory diseases such as encephalitis or meningitis, craniocerebral trauma or spinal cord injury), or peripheral nervous system injury or lesions within 6 months before signing the informed consent;
10. History of myopathy/myalgia, or susceptibility to myopathy/rhabdomyolysis (e.g., family history of hereditary myopathy, previous use of HMG-CoA reductase inhibitors in combination with fibrates, etc.);
11. Presenting with hypothyroidism, defined as marked TSH elevations (usually > 1.5 ULN) associated with decreases in free T4 (FT4) ;
12. Patients with a history of drug abuse, drug abuse and alcoholism (tolerance, withdrawal, impaired control of drinking behavior) in the past 1 year;
13. Participation in another interventional clinical investigator within 1 month prior to informed consent;
14. Patients who, in the opinion of the investigator, are not suitable for this study.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2026-06-16 (Estimated); Study Completion 2026-11-14 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in IIEF-EF (Questions 1-5 and 15 in the IIEF scale) score at Week 13 visit; | 12 weeks
Change From Baseline in Carotid Artery Intima-media Thickness (IMT) by Peripheral Ultrasound at Week 13 Visit. | 12 weeks

SECONDARY OUTCOMES:
Adverse event (AE)/serious adverse event (SAE); | 16 weeks

IPD SHARING:
Plan to Share IPD: No